CLINICAL TRIAL: NCT03458442
Title: China OLIMPICS: China Ophthalmic Learning and Improvement Initiative in Cataract Surgery Trial, an Education-Intervention Randomized Control Study
Brief Title: China OLIMPICS: China Ophthalmic Learning and Improvement Initiative in Cataract Surgery Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Congdon Nathan, Professor of Preventative Ophthalmology, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: China OLIMPICS* Trial
Record Dates: First submitted 2017-10-07; First posted 2018-03-08 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2019-04

CONDITIONS: Cataract
Keywords: education; developing country; developing countries; low-and middle-income country; low-and middle-income countries; surgical training; blindness; china; simulation; model
MeSH Terms: conditions — Cataract; Blindness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Standard surgical training + simulation-based surgical training
  Interventions: Other: Simulation-based surgical training; Other: Standard surgical training
- Control Arm (Active Comparator): Standard surgical training
  Interventions: Other: Standard surgical training

INTERVENTIONS:
Other: Simulation-based surgical training — Those in the intervention group will be introduced to a variety of simulation-based surgical training techniques. Specifically, this will involve breaking down the SICS cataract surgery procedure into stages, and practicing each stage repeatedly using simulation. This sustained deliberate practice will be integrated into the six-week course, as an enhancement to the course, and not as a replacement of any part of the educational content. Within the last three weeks of the course, 'intervention' arm participants will be introduced to the artificial eyes, the Simulation-OSSCAR rubric, and be provided with ongoing feedback.
  All participants in both intervention and control arms will undertake the six-week Orbis-COS training course.
  Arms: Intervention Arm
Other: Standard surgical training — Standard surgical training (without bespoke training scheme using simulation and model eye). All participants in both intervention and control arms will undertake the existing six-week Orbis-COS training course, which includes 2-4 weeks of didactic lectures, surgical observation, and wet lab training with a minimum of 50 pig eye wet lab simulations per trainee. After observed mastery of wet lab pig eyes, trainees then perform hands-on training in county level hospitals. The hands-on training pairs a surgeon from the training centre to mentor the trainee through a minimum of 30 assisted surgeries and 50 independent surgeries under supervision.

SUMMARY:
This is a prospective, investigator-masked randomised controlled education-intervention trial of intense simulation-based surgical education plus conventional training versus a current six-week standard training course. The aim is to investigate whether the addition of simulation-based surgical education to standard training improves competence and surgical outcomes. All participants in the study will receive the educational intervention of the six-week Orbis-COS course. The intervention groups will receive this training and an additional element of learning and sustained deliberate practice using model eyes and simulation.

DETAILED DESCRIPTION:
Project Description:

The leading cause of blindness in China and the world is un-operated cataract. Despite notable efforts on the part of the Chinese government, China's cataract surgical rate (1400/million/year in 2015) remains behind that of many of its poorer neighbours, such as India (6500) and Vietnam (2250). An important reason is the unavailability of trained surgeons: though China has over 36,000 ophthalmologists, only a third are capable of performing independent cataract surgery. This shortfall is due in large part to lack of hands-on training opportunities. A recent survey of residents at China's top-ranked resident training programs found that the median number of independent cataract surgeries performed was actually zero. The problem persists after formal training is completed: <5% of cataract surgeries are performed by doctors aged 24-43 years. The problem is particularly acute in rural areas, where hands-on training opportunities for young ophthalmic surgeons are even rarer. One reason is safety concerns on the part of patients and senior doctors in entrusting operations to young surgeons.

New training models for cataract surgery are needed which can safely and efficiently support trainees during the transition from novice to competent surgeon. Simulation-based surgical training, using high-fidelity, inexpensive, re-usable model eyes have been successfully piloted. The investigators now propose to carry out a randomized trial comparing training using these model eyes with traditional techniques, to study the impact on quality of surgery (assessed by masked grading of videos using the ICO OSCAR system), visual acuity and cost-utility outcomes.

The investigators research will reduce expenses by piggybacking on an on-going collaborative program between Orbis International, the Chinese MOH, Chinese National Blindness Prevention Committee and Tongren Hosptal (one of China's largest and best-respected eye hospitals), which will train 120 rural cataract surgeons at 60 county hospitals in 6 provinces. The study's collaboration involves internationally-respected vision research teams at ICEH, Queen's University Belfast and Tongren, while offering opportunities for scale-up and engagement with Chinese policy makers at the highest level.

A successful trial proving the training benefits of inexpensive model eyes will make a unique contribution to building the capacity to manage China's leading cause of blindness, thus furthering the aims of SightFirst and the Chinese Ministry of Health, while improving the lives of Chinese people dwelling in low-resource areas.

ELIGIBILITY:
Inclusion Criteria:

* Surgeon Inclusion Criteria:

  * <20 complete SICS cases performed lifetime
  * Completed ophthalmic training or in residency training with license to perform surgery
  * Will have opportunity to carry out independent SICS surgery after training
* Patient Enrolment Criteria:

  * Cataract in one or both eyes felt to be visually significant in the opinion of the operating ophthalmologist.

Exclusion Criteria:

* Surgeon Exclusion Criteria:

  * Already capable of performing independent intra-ocular surgery of any kind
  * No opportunity to perform cataract surgery after training.
* Patient Exclusion Criteria:

  * Fellow eye has an irreversible cause of visual impairment
  * Any prior ophthalmic surgery in the proposed operative eye
  * Any co-morbid condition in the operative eye likely to impact post-operative visual acuity negatively (conditions only detected on post-operative examination would also lead to retrospective exclusion.)

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Surgical Skill - ICO OSCAR Score | First 10 successive independent surgeries after training--expected within 6 months after completion of training
  Mean video grade of first 10 successive supervised or assisted SICS cases (with patient consent) for each trainee surgeon, using ICO-OSCAR. Two approaches to determine mean video grade will be employed to account for variation in the number of surgical steps performed by trainees.
  Both approaches are equally significant for determining main outcome, differing solely in number of steps graded.
  * Mean video grade across all surgical steps of first 10 supervised SICS cases for each trainee, using ICO-OSCAR. This approach assigns a score 0 for steps not performed.
  * Mean video grade across all trainee-completed steps of first 10 supervised SICS cases for each trainee, using ICO-OSCAR. This approach takes into consideration mentors' teaching styles.
  The graders are masked to surgeon/patient identity, using a file-sharing platform to transfer videos to graders and collate grading information. These are the first 10/30 cases completed under STEER trainer supervision.

SECONDARY OUTCOMES:
Post-operative Presenting Visual Acuity | Post-operative day #1
  Mean presenting logMAR visual acuity, on post-operative day #1 of 10 successive cases per surgeon (measured using the BOOST [Better Operative Outcome Software Tool] application.
Post-operative Improvement in Visual Acuity | Post-operative day #1
  Mean improvement in lines of visual acuity, on post-operative day #1 of 10 successive cases per surgeon (measured using the BOOST [Better Operative Outcome Software Tool] application.
Cost per trainee | After conclusion of study activity--calculated up to 1 month after data from final surgery collected
  Cost per trainee in each wing

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD, MPH, Principal Investigator — Zongshan Ophthalmic Center; William Dean, FRCO MBChB, Principal Investigator — London School of Hygiene and Tropical Medicine; Ningli Wang, Principal Investigator — Tongren Hospital
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murthy G, Gupta SK, John N, Vashist P. Current status of cataract blindness and Vision 2020: the right to sight initiative in India. Indian J Ophthalmol. 2008 Nov-Dec;56(6):489-94. doi: 10.4103/0301-4738.42774. PMID 18974520
- [Background] Young AL, Jhanji V, Liang Y, Congdon N, Chow S, Wang F, Zhang X, Man X, Yang M, Lin Z, Yuen HG, Lam DS. A survey of perceived training differences between ophthalmology residents in Hong Kong and China. BMC Med Educ. 2015 Sep 28;15:158. doi: 10.1186/s12909-015-0440-0. PMID 26415932
- [Background] Resnikoff S, Felch W, Gauthier TM, Spivey B. The number of ophthalmologists in practice and training worldwide: a growing gap despite more than 200,000 practitioners. Br J Ophthalmol. 2012 Jun;96(6):783-7. doi: 10.1136/bjophthalmol-2011-301378. Epub 2012 Mar 26. PMID 22452836
- [Background] Golnik C, Beaver H, Gauba V, Lee AG, Mayorga E, Palis G, Saleh GM. Development of a new valid, reliable, and internationally applicable assessment tool of residents' competence in ophthalmic surgery (an American Ophthalmological Society thesis). Trans Am Ophthalmol Soc. 2013 Sep;111:24-33. PMID 24072944

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT03458442/Prot_SAP_ICF_001.pdf